CLINICAL TRIAL: NCT03838055
Title: Sentinel Lymph Node Detection in Endometrial Cancer: A Consolidation Study
Brief Title: Sentinel Node Detection in Endometrial Cancer: A Consolidation Study on Detection Rates of Metastatic Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RegionSkaneKKLund3
Record Dates: First submitted 2018-12-21; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Sentinel Lymph Node; Endometrial Cancer; Lymphedema
MeSH Terms: conditions — Endometrial Neoplasms; Lymphedema

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SLN only (Experimental): Pelvic SLN's defined by ICG injected cervically
  Interventions: Procedure: Injection of tracer ( ICG) and detection of sentinel lymph nodes

INTERVENTIONS:
Procedure: Injection of tracer ( ICG) and detection of sentinel lymph nodes — Pelvic SLN's defined by ICG injected cervically

SUMMARY:
Evaluation of removal of Sentinel lymph nodes only for detection of pelvic lymph node metastases in high risk and low risk endometrial cancer.

DETAILED DESCRIPTION:
Consecutive patients with- and low risk endometrial cancer will be approached for eligibility for inclusion in a study evaluating the detection rates of pelvic metastatic disease by detection and removal of Sentinel lymph nodes only, i.e with no further lymphadenectomy.

A re-staging will be performed in case of metastatic Sentinel lymph nodes to guide adjuvant treatment.

The detection rate will be evaluated from a non-inferiority perspective against the expected rate of nodal metastases based on detailed final histological data.

Adverse events related the intervention ( Injection of tracer (ICG) and removal of sentinel nodes), time for the intervention, and an objective evaluation of lymphatic complications (lymphoedema) will be performed in addition to the use of a validated lymphoedema QOL questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Women of age 18 years and older at the time of informed consent.
* Women with a pathologically proven endometrial carcinoma of any histologic subtype or grade, clinically stage I-II planned for primary surgery
* A uterine size allowing minimally invasive surgery
* Women must be able to understand and sign an informed consent in Swedish language.
* Absence of any exclusion criteria

Exclusion Criteria:

* Non consenting patients
* Ongoing pregnancy
* Inability to understand written and/or oral study information
* WHO performance status or conditions contraindicating adjuvant oncological treatment (WHO III or more)
* Previous lower limb lymphedema ( only for the lymphedema part of study)
* Evidence of locally advanced disease or intraabdominal/distant metastases at preoperative CT, MRI or ultrasonography.
* Surgical contraindication to a laparoscopic approach or lymphadenectomy at surgeons discretion.
* Anesthesiologic contraindication to a laparoscopic approach at the anesthetist's discretion
* Allergy to Iodine
* Patients with a known liver disease
* Patients with a bleeding disorder or mandatory antithrombotic treatment.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 362 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate of pelvic metastatic disease in endometrial cancer | 3 years from start inclusion with an interim analysis after 150 patients
  The detection rate will be evaluated from a non-inferiority perspective based on a null-hypothesis of 4% less than an expected rate of 12% nodal metastases
Operative time used for the study intervention ( injection of ICG and identification and removal of sentinel lymph nodes | 3 years from start inclusion
  Exact measurements of time allocated for the SLN procedure as such.

SECONDARY OUTCOMES:
Incidence of lymphedema after removal of sentinel lymph nodes | 4 years including at least one year follow up
  Objective measurement lymphedema defined by of leg volume before and after surgery
intraoperative adverse events associated with the study intervention | 3 years from start inclusion or after 150 patients if study stopped at interim analysis
  Detailed registration of adverse events associated with the SLN procedure as such

CONTACTS AND LOCATIONS:
Overall Officials: Jan Persson, Ass Prof, Principal Investigator — RegionSkane, department of OB&G, Skåne university hospital, Lund
Locations (1):
- Department of Gynecology and Obstetrics, Lund, Sweden

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT03838055/Prot_SAP_000.pdf